CLINICAL TRIAL: NCT03975348
Title: Evaluation of Ventilation Distribution After Bariatric Surgery - High Flow Nasal Cannulas Versus Continuous Positive Airway Pressure
Brief Title: Ventilation Distribution After Bariatric Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Trieste (Other)
Responsible Party: Principal Investigator, Lucia Comuzzi, Principal investigator, University of Trieste
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 123/2018
Record Dates: First submitted 2019-05-03; First posted 2019-06-05 (Actual); Last update posted 2020-07-30 (Actual); Status verified 2020-07

CONDITIONS: Bariatric Surgery Candidate; Atelectasis, Postoperative Pulmonary
Keywords: High flow nasal cannula; Bariatric surgery; Postoperative atelectasis; Electrical impedance tomography
MeSH Terms: conditions — Pulmonary Atelectasis | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (10):
- Baseline conventional facemask (Other): The patients will receive oxygen therapy through conventional facemask for 10 minutes
  Interventions: Device: Facemask
- HFNC 40 L/min up (Experimental): The patients will receive oxygen/air mixture through high flow nasal cannula at incremental, then decremental flows, starting at 40 L/min for 10 minutes
  Interventions: Device: High flow nasal cannula
- HFNC 60 L/min up (Experimental): High flow nasal cannula at 60 L/min for 10 minutes
  Interventions: Device: High flow nasal cannula
- HFNC 80 L/min up (Experimental): High flow nasal cannula at 80 L/min for 10 minutes
  Interventions: Device: High flow nasal cannula
- HFNC 100 L/min (Experimental): High flow nasal cannula at 100 L/min for 10 minutes
  Interventions: Device: High flow nasal cannula
- HFNC 80 L/min down (Experimental): High flow nasal cannula at 80 L/min for 10 minutes
  Interventions: Device: High flow nasal cannula
- HFNC 60 L/min down (Experimental): High flow nasal cannula at 60 L/min for 10 minutes
  Interventions: Device: High flow nasal cannula
- HFNC 40 L/min down (Experimental): High flow nasal cannula at 40 L/min for 10 minutes
  Interventions: Device: High flow nasal cannula
- Washout conventional facemask (Other): Again, the patients will receive oxygen therapy through conventional facemask for 10 minutes, to reduce the influence of HFNC on CPAP therapy
  Interventions: Device: Facemask
- CPAP (Active Comparator): The patients will receive CPAP at 10 cmH2O for 10 minutes
  Interventions: Device: Continuous positive airway pressure

INTERVENTIONS:
Device: High flow nasal cannula — High flow of warm and humidified oxygen/air mixture delivered through nasal cannula
  Arms: HFNC 100 L/min; HFNC 40 L/min down; HFNC 40 L/min up; HFNC 60 L/min down; HFNC 60 L/min up; HFNC 80 L/min down; HFNC 80 L/min up
Device: Continuous positive airway pressure — Positive airway pressure applied through a sealed face mask
  Arms: CPAP
Device: Facemask — Oxygen therapy through a conventional facemask
  Arms: Baseline conventional facemask; Washout conventional facemask

SUMMARY:
Obese patients have an increased risk of developing post-operative respiratory complications due to their comorbidities. They have a restrictive ventilatory defect with reduction of lung volumes and expiratory flow limitation, higher airway resistance and collapsibility of the upper respiratory tract. These abnormalities are worsened by general anesthesia and opioid administration. It has been proved that oxygen therapy with HFNC (high flow nasal cannula) increases lung volumes through a continuous positive airway pressure (CPAP)-effect. This also improves gas exchange and decreases anatomical dead space. At the present time, CPAP represents the gold standard for the prevention of postoperative pulmonary complications. The purpose of this study is to evaluate lung ventilation, gas exchange and comfort with HFNC compared with CPAP during the post-operative period in patients who undergo laparoscopic bariatric surgery.

DETAILED DESCRIPTION:
Immediately after bariatric surgery, patients will follow a pre-determined schedule of oxygen therapy with conventional facemask (from the beginning to minute 10), HFNC (with a flow of 40 L/min from minute 11 to 20, 60 L/min from minute 21to 30, 80 L/min from minute 31 to 40, 100 L/min from minute 41 to 50, 80 L/min from minute 51 to 60, 60 L/min from minute 61 to 70, 40 L/min from minute 71 to 80), conventional facemask again (washout, from minute 81 to 90) and CPAP (10 cmH2O, from minute 91 to 100). Lung ventilation will be evaluated with electrical impedance tomography (EIT), which measures thoracic impedance variations related to changes in lung aeration. At the end of each 10 minutes-period the following data will be collected: electrical impedance tomography data (to calculate the global inhomogeneity index, Δ end-expiratory lung impedance and tidal impedance variation), hemodynamic parameters, respiratory rate, SpO2, pain (numerical rating scale), level of sedation (Ramsey score) and patient comfort (modified Borg scale). An arterial blood gas will be collected at the end of the following steps: baseline facemask, HFNC 40 and 100 L/min, washout facemask and CPAP. Data about anesthetic/analgesic drugs and ventilation parameters will also be collected.

ELIGIBILITY:
Inclusion Criteria:

* Patient's consent to the trial
* Candidate to laparoscopic bariatric surgery (sleeve gastrectomy or Roux-en-Y gastric bypass)
* BMI 35-50 kg/m2
* ASA class 1-3

Exclusion Criteria:

* Obesity hypoventilation syndrome
* Contraindication to EIT (e.g. implantable cardioverter-defibrillator)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2019-04-15 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Change of global inhomogeneity index | The data needed to calculate the index will be collected at minute 10, 20, 30, 40, 50, 60, 70, 80, 90 and 100 (i.e. at the end of every step of oxygen therapy). The values obtained will then all be compared each other.
  This parameter, calculated from data collected with EIT, evaluates lung ventilation distribution. To calculate this index, the median value of regional impedance changes from ventilated regions within the tidal image has to be computed, then the sum of differences between the median and every pixel value needs to be calculated, and the result must be normalised by the sum of impedance values within the lung area. The minimum value of the index is 0 and corresponds to homogeneous ventilation, whereas the maximum value is 1 and corresponds to inhomogeneous ventilation (in this context likely due to atelectasis).

SECONDARY OUTCOMES:
Change of Δ end expiratory lung impedance (ΔEELI) | The data will be collected at minute 10, 20, 30, 40, 50, 60, 70, 80, 90 and 100 (i.e. at the end of every step of oxygen therapy). The values obtained will then all be compared each other.
  The parameter, measured with EIT, expresses deviations of the regional end-expiratory lung impedance in relation to the global tidal impedance variation. ΔEELI closely correlates with changes of end-expiratory lung volume of the EIT sensitivity region.
Change of tidal impedance variation | The data will be collected at minute 10, 20, 30, 40, 50, 60, 70, 80, 90 and 100 (i.e. at the end of every step of oxygen therapy). The values obtained will then all be compared each other.
  This parameter, measured with EIT, corresponds to the difference between end-expiratory and end-inspiratory lung impedance and is related to tidal volume. It will be expressed in units, where one unit corresponds to the tidal impedance variation of the patient breathing with baseline conventional facemask.
Change of oxygenation | The blood gas analysis will be performed at minute 10, 20, 50, 90 and 100. The values will then all be compared each other.
  Oxygen arterial partial pressure
Change of carbon dioxide | The blood gas analysis will be performed at minute 10, 20, 50, 90 and 100. The values will then all be compared each other.
  Carbon dioxide arterial partial pressure
Change of pH | The blood gas analysis will be performed at minute 10, 20, 50, 90 and 100. The values will then all be compared each other.
  Arterial pH
Change of respiratory rate | The parameter will be collected at minute 10, 20, 30, 40, 50, 60, 70, 80, 90 and 100 (i.e. at the end of every step of oxygen therapy). The values obtained will then all be compared each other.
  Respiratory rate
Change of patient's comfort: modified Borg dyspnea scale | The parameter will be collected at minute 10, 20, 30, 40, 50, 60, 70, 80, 90 and 100 (i.e. at the end of every step of oxygen therapy). The values obtained will then all be compared each other.
  Comfort related to the oxygen therapy will be evaluated with the modified Borg dyspnea scale (0: nothing at all, 0.5: very, very slight, 1: very slight, 2: slight, 3: moderate, 4: somewhat severe, 5: severe, 6, 7: very severe, 8, 9: very, very severe - almost maximal, 10: maximal)

CONTACTS AND LOCATIONS:
Overall Officials: Lucia Comuzzi, Principal Investigator — Azienda Sanitaria Universitaria Integrata di Trieste
Locations (1):
- Azienda Sanitaria Universitaria Integrata di Trieste, Trieste, Italy

IPD SHARING:
Plan to Share IPD: No